CLINICAL TRIAL: NCT06373419
Title: Thulium Fiber Laser (TFL) Versus MOSES Holmium Laser in the En-bloc Resection of Bladder Tumors: A Randomized Controlled Clinical Study
Brief Title: TFL vs MOSES Holmium Laser in the En-bloc Resection of Bladder Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Principal Investigator, Ahmed Zakaria Ahmed, Urologist, Thunder Bay Regional Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-1007
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Urolithiasis of Bladder
MeSH Terms: conditions — Urinary Bladder Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium Fibre Laser (Active Comparator): Participants randomized to this arm will undergo bladder resection using the TFL laser
  Interventions: Device: TFL
- MOSES Holmonium (Active Comparator): Participants randomized to this arm will undergo bladder resection using the MOSES holmium laser.
  Interventions: Device: MOSES holmium laser

INTERVENTIONS:
Device: TFL — Participant undergoing bladder tumour resection that has been randomized to this arm.
  Arms: Thulium Fibre Laser
Device: MOSES holmium laser — Participant undergoing bladder tumour resection that has been randomized to this arm.
  Arms: MOSES Holmonium

SUMMARY:
The goal of this randomized clinical trial is to determine if there is difference in pathological and clinical outcomes between MOSES and TFL in the transurethral laser enucleation of bladder tumors.

The main question it aims to answer is:

Is there a difference in pathological and clinical outcomes between MOSES Holmium and Thulium Fiber Laser (TFL) in the transurethral laser enucleation of bladder tumors?

Participants will randomized to either TFL of MOSES arm for their bladder resection procedure.

DETAILED DESCRIPTION:
An estimated 12,500 Canadians are diagnosed with bladder cancer each year. Diagnosis and treatment involve transurethral (through the urethra) resection of tumor or tissue called the TURBT procedure. This procedure yields excellent results and minimal morbidity and mortality but has a high recurrence rate, difficulties in the pathologic interpretation of the specimen (due to cautery effect), and procedure-related complications (excessive bleeding, bladder perforation, bowel injury, and inadvertent extensive injury to urethra) that may delay treatments such as chemotherapy which would further impact oncologic outcomes. With the advancement of technology, new methods of transurethral tumor removal have emerged, such as the use of laser energy. Using laser energy, the tumour is resected in one piece, whereas the TURBT approach requires breaking the tumor into pieces. This allows for better pathology analysis that can determine treatment pathways for the patient, as well as reduces the risk of complications. The standard lasers used have been the MOSES Holmium laser and the Thulium Fiber Laser (TFL).

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age at the time of enrollment.
2. Patients presented with visual criteria suggesting bladder tumor by outpatient cystoscopy will be legible for inclusion.

Exclusion Criteria:

1. Tumors deemed not eligible for laser resection as determined by the Urologist e.g. obvious muscle-invasive or metastatic at presentation
2. Synchronous either urethral tumors or upper urinary tract tumor
3. History of Carcinoma in situ
4. Contracted bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Presence of muscularis propria | 1 day post-procesure
  Presence of muscularis propria (bladder muscle cells) in the pathology sample of the bladder tumour
Incidence of inconclusive pathology | 1 day post-procedure
  Incidence of inconclusive pathology due to specimen artifact

SECONDARY OUTCOMES:
Tumor-free rate (TFR) | 6 to 12 weeks post-procedure
  As per the follow-up cystoscopy, TFR is defined as the absence of any residual tumor detectable by cystoscopy.
Total operative time | Intraoperative
  In minutes measured from anesthesia induction until placement of the urethral catheter
Total procedural time | Intraoperative
  In minutes, measured from the time the cystoscope sheath is inserted into the participant to the time the cystoscope has been removed
Number of recurrences | 12 weeks post-procedure
  Defined as any tumor detection by follow-up cystoscopy after the initial resection
Total blood loss | 6 hours post-procedure
  Defined as a drop in hemoglobin level from pre-op
Rate of complications | 4 weeks post-procedure
  Percentage of participants with post-operative complications
Number of inconclusive pathology | 1 day post-procedure
  Number of inconclusive pathology due to thermal effect artifact.
Lasing time | Intraoperative
  In minutes, defined as the time the laser was in use, not including pedal pauses
Total energy used | Intraoperative
  Measured in kilojoules
Frequency and severity of peri-operative complications | Intraoperative
  Reported according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Z Ahmed, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No